CLINICAL TRIAL: NCT05632653
Title: Percutaneous Coronary Intervention in Patients with Chronic Total Occlusion of Coronary Arteries and Heart Failure.
Brief Title: CTO-PCI in Heart Failure Patients
Acronym: CTO-HF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: Herzzentrum Lahr (Unknown); IHF GmbH - Institut für Herzinfarktforschung (Other)
Responsible Party: Principal Investigator, Michael Behnes, Prof. Dr. med., Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01012022-MA
Record Dates: First submitted 2022-01-27; First posted 2022-11-30 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Coronary Artery Disease; Chronic Total Occlusion; Heart Failure
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTO-PCI (Experimental)
  Interventions: Procedure: CTO-PCI
- non-CTO-PCI (No Intervention)

INTERVENTIONS:
Procedure: CTO-PCI — Percutaneous coronary intervention (PCI) of a coronary chronic total occlusion (CTO) (CTO-PCI) in patients with systolic heart failure (LVEF <50%).
  Arms: CTO-PCI

SUMMARY:
The study investigates wheather CTO-PCI improves survival and heart failure related rehospitalization compared to optimal medical therapy (OMT). This hypothesis will be investigated within a large-scaled international, representative, prospective, randomized, controlled, open-label, event-driven, multicentre trial (trial acronym: CTO - Heart Failure) recruiting patients with planned CTO-PCI.

DETAILED DESCRIPTION:
Coronary artery disease (CAD) is the most common cause of heart failure and death worldwide. Beside non-occlusive coronary arterial stenoses, 25% of CAD patients have a so called chronic total occlusion (CTO) at one out of three main coronary arteries. CTO are often left untreated by physicians over many years due to lack of knowledge of its prognostic relevance and due to be too challenging and risky for the interventional cardiologist, particularly in the presence of severe comorbidities such as heart failure. By development of new interventional devices, techniques and algorithms, CTO can be revascularized in more than 90% with low complication rates. Per se, a patient suffering from comorbid heart failure caused by CAD including a CTO is often regarded as inoperable for heart surgery by coronary artery bypass grafting (CABG). Therefore, the only causal alternative therapy represents the less-invasive interventional revascularization of the CTO by percutaneous coronary intervention (PCI). Until now, the prognostic impact of CTO-PCI has never been proven. Our recent work has outlined the beneficial impact of CTO-PCI to improve both left ventricular cardiac function and cardiopulmonary exercise capacity in patients with heart failure. Our objective is to understand whether CTO-PCI improves survival and heart failure related rehospitalization compared to optimal medical therapy (OMT). This hypothesis will be investigated within a large-scaled representative, prospective, randomized, controlled, open-label, event-driven, multicentre trial (trial acronym: CTO - Heart Failure) recruiting patients with planned CTO-PCI. The CTO Heart Failure aims to deliver evidence whether CTO-PCI might become a prognostically relevant established therapeutic option for patients with systolic heart failure.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Presence of at least one CTO located at the proximal to midpart of left artery descending (LAD), or at proximal left circumflex (LCX), or at proximal to midpart LCX in left dominant system, or at proximal to distal right coronary artery (RCA).
* LVEF <50% (assessed within 6 weeks prior to enrolment by transthoracic echocardiography (TTE) (Simpson biplane method) or cardiac magnetic resonance imaging (cMRI).
* In patients with multivessel disease (MVD) and Syntax I score ≥ 22, and all patients with type 2 diabetes and coronary 3 vessel disease, a heart team decision favouring CTO-PCI is needed.
* Mandatory baseline imaging assessment (assessed within 6 weeks prior to enrolment):
* TTE: Normal wall motion or hypokinesia in the CTO-territory.
* In case of severe hypokinesia, akinesia or dyskinesia a viability testing with cMRI or myocardial scintigraphy (MS) indicating at least 50% of viability in the CTO territory (mandatory only in the presence of akinesia in the CTO-territory assessed by prior TTE) prior to PCI is mandatory.
* Symptoms including dyspnea (according to the New York Heart Association (NYHA), classes II-III) or angina pectoris (according to Canadian Cardiovascular Society (CCS), classes II-IV).
* In the absence of symptoms evidence of myocardial ischemia of at least 10% is needed being assessed by invasive or non-invasive imaging, such as stress-MRI, PET-CT-scan, myocardial scintigraphy, stress-echocardiography

Exclusion Criteria:

* Age <18 and >90 years.
* Akinesia or dyskinesia assessed by TTE plus subendocardial late gadolinium enhancement of >50% assessed by cMRI or MS in the CTO-territory or any evidence of transmural scarring of the CTO-territory (i.e. 100%).
* Presence of terminal kidney disease with need for renal replacement therapy.
* Severe chronic kidney disease (defined as GFR < 25 ml/min).
* Type I myocardial infarction (ST segment elevation or non-ST segment elevation myocardial infarction (STEMI or NSTEMI)) related to critical arteriosclerosis < 30 days.
* End-stage heart failure (defined by constant administration of intravenous inotropes, use of prolonged assist devices (more than 5 days), listing for high urgent cardiac transplantation).
* Cardiogenic shock (< 30 days).
* Heart team decision favoring CABG surgery (in the presence of coronary multivessel disease with intermediate to high SYNTAX I score).
* Grade II-III heart valve disorders requiring interventional or surgical treatment within 3 months.
* Right-sided heart failure with echocardiographic evidence of severe right ventricular dysfunction.
* COPD requiring long-term oxygen therapy.
* Non-cardiac comorbidity with life expectancy < 12 months.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 783 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2030-03 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Composite of all-cause mortality or heart failure related rehospitalization. | up to 3 years
  Heart failure related rehospitalization is defined as a rehospitalization due to worsening heart failure requiring intravenous therapy as the primary cause, or as a result of another cause but associated with worsening heart failure at the time of admission, or as a result of another cause but complicated by worsening heart failure during its course

SECONDARY OUTCOMES:
Canadian cardiovascular society (CCS) class | up to 3 years
  angina pectoris
All-cause mortality. | up to 3 years
Heart failure related rehospitalization. | up to 3 years
MACCE | up to 3 years
  MACCE are defined as the composite of all-cause death, myocardial infarction (type I and II), any further type of coronary revascularization (i.e. PCI or CABG) based on functional invasive assessment by fractional flow reserve (FFR) or instantaneous wave-free ratio (iFR), and stroke.
Number of participanty with rehospitalization due to cardiac diseases beyond heart failure. | up to 3 years
assessment of quality of life | up to 3 years
  Seattle angina questionnaire (SAQ) (0-100; 75-100 normal).
cost effectivenes | up to 3 years
  direct and indirect health care related costs
Re-assessment of LVEF | up to 3 years
New York Heart association (NYHA) class | up to 36 months
  dyspnea

CONTACTS AND LOCATIONS:
Overall Officials: Michael Behnes, Prof. Dr., Principal Investigator — Universitätsmedizin Mannheim; Kambis Mashayekhi, PD Dr., Study Director — MEDICLIN Herzzentrum Lahr

IPD SHARING:
Plan to Share IPD: No